CLINICAL TRIAL: NCT02148653
Title: Efficacy of an Antiinflammatory Diet as Modulator of Cardiometabolic Risk and Body Weight in Healthy Overweight Subjects: Studies of Mechanisms Involving Metabolomics and Gut Microbiota Mapping
Brief Title: An Antiinflammatory Diet as Modulator of Cardiometabolic Risk and Body Weight in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Vinnova (Other Government)
Responsible Party: Principal Investigator, Juscelino Tovar, Project Manager, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AFC-JT-MFD
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Overweight
Keywords: Cardiometabolic risk; Diet; Dietary prevention; Functional diet; Functional foods; Metabolic Syndrome; Overweight
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifunctional diet (MFD) (Experimental): Subjects eat a diet designed according to the Nordic Nutrition Recommendations with the addition of important amounts of various functional food concepts: Low GI and GI-modulating food items; Natural antioxidant-rich items, Long chain omega-3 fatty acid-rich fish; Betaglucan-rich barley and oat food/drinks; Cholesterol-modulating foods.
  Interventions: Other: Multifunctional diet (MFD)
- Control diet (Experimental): Subjects eat a diet designed according to the Nordic Nutrition Recommendations but lacking the functional items included in the MFD.
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Multifunctional diet (MFD) — A mixed diet containing multiple functional foods/concepts with the ability to modulate blood lipid levels, glycemia, insulinemia and prothrombotic status.
  Arms: Multifunctional diet (MFD)
Other: Control diet — A nutritionally well formulated diet that excludes the functional food items present in the MFD.
  Arms: Control diet

SUMMARY:
Main scientific question:

A previous intervention with an anti-inflammatory multifunctional dietary portfolio (MFD) showed remarkable reductions in cardiometabolic (CM) risk markers compared with a well-designed control diet. The study was performed under weight maintenance conditions in healthy subjects in a 4w crossover design (Tovar et al., 2012). MFD consumption also resulted in improved cognitive performance after 4 weeks (Nilsson et al., 2013).

The present project will further study the preventive potential of MFD, using its unique properties for identification of new biomarkers and to evaluate the potential role of alterations in the gut microbiota. MFD will be tested in healthy at risk subjects in a randomized parallel design in an eight-week intervention with the test or control diet, respectively, allowing for weight loss. Assessment of standard anthropometric/biochemical markers of CM risk, metabolomics analysis and appetite regulating hormone evaluation are also planned. Associations between the gut microbiota composition and measures of CM risk are also included. The project provides unique opportunities to identify mechanisms for the metabolic impact of MFD, for further exploitation in innovative food and/or dietary concepts.

Central hypothesis:

The CM-preventive potential of MFD may be boosted in a medium-term trial under conditions allowing for body weight reduction. Expected additional benefits may be recorded as reduced values for conventional CM-related parameters, markers of modified gut microbiota composition and specific changes in blood metabolite profiles.

Objectives:

* To further improve the effect of MFD on biochemical/anthropometric CM risk markers in healthy subjects by administering the diet under conditions allowing for weight reduction.
* To identify MFD-related changes in the gut microbiota associated with improved CM risk markers.
* To assess MFD-related modification in metabolic pathways, studied with a metabolomics approach, and to correlate them with conventional clinical outcomes, aiming to identify new markers of altered metabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Normal fasting blood glucose (max 6.1 mmol /l)
* BMI between 25 and 32 Kg/m2

Exclusion Criteria:

* treatment for hypercholesterolemia
* treatment for hypertension
* history of cardiovascular complications

Ages: 50 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in LDL cholesterol after each dietary period | Time 0 and after week 8
  Start and End of the intervention arm

SECONDARY OUTCOMES:
Change from baseline in body weight after each dietary period | Week 0 and after 8 weeks
  Start and End of the intervention arm

OTHER OUTCOMES:
Change from baseline in circulating triglycerides | Week 0 and after 8 weeks
  Start and End of the intervention arm
Change from base line in the diversity of gut microbiota | Week 0 and after 8 weeks
  Start and End of the intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Juscelino Tovar, PhD, Study Chair — Antidiabetic Food Centre & Functional Food Science Centre. Lund University
Locations (1):
- Functional Food Science Centre. Lund University Medicon Village, Lund, Sweden

REFERENCES:
- [Background] Tovar J, Nilsson A, Johansson M, Ekesbo R, Aberg AM, Johansson U, Bjorck I. A diet based on multiple functional concepts improves cardiometabolic risk parameters in healthy subjects. Nutr Metab (Lond). 2012 Apr 2;9:29. doi: 10.1186/1743-7075-9-29. PMID 22472183
- [Background] Nilsson A, Tovar J, Johansson M, Radeborg K, Bjorck I. A diet based on multiple functional concepts improves cognitive performance in healthy subjects. Nutr Metab (Lond). 2013 Jul 15;10:49. doi: 10.1186/1743-7075-10-49. eCollection 2013. PMID 23855966
- [Result] Tovar J, Johansson M, Bjorck I. A multifunctional diet improves cardiometabolic-related biomarkers independently of weight changes: an 8-week randomized controlled intervention in healthy overweight and obese subjects. Eur J Nutr. 2016 Oct;55(7):2295-306. doi: 10.1007/s00394-015-1039-2. Epub 2015 Sep 14. PMID 26370118
- [Derived] Arroyo CB, Ocariz MG, Rogova O, Al-Majdoub M, Bjorck I, Tovar J, Spegel P. A randomized trial involving a multifunctional diet reveals systematic lipid remodeling and improvements in cardiometabolic risk factors in middle aged to aged adults. Front Nutr. 2023 Sep 14;10:1236153. doi: 10.3389/fnut.2023.1236153. eCollection 2023. PMID 37781111
- [Derived] Marungruang N, Tovar J, Bjorck I, Hallenius FF. Improvement in cardiometabolic risk markers following a multifunctional diet is associated with gut microbial taxa in healthy overweight and obese subjects. Eur J Nutr. 2018 Dec;57(8):2927-2936. doi: 10.1007/s00394-017-1563-3. Epub 2017 Nov 2. PMID 29098426